CLINICAL TRIAL: NCT02744963
Title: Carefully seLected and Easily Accessible at No Charge Medications
Acronym: CLEAN-Meds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: The Ontario Spor Support Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-114
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Medication Adherence; Inappropriate Prescribing; Diabetes; Hypertension
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Free and convenient medicine access (Experimental): Free access to a list of essential medicines. Medicines are either mailed to the patient or dispensed at the point of care.
  Interventions: Other: Free and convenient medicine access
- Usual medicine access (No Intervention): Usual access to medicines.

INTERVENTIONS:
Other: Free and convenient medicine access
  Arms: Free and convenient medicine access

SUMMARY:
This trial evaluates the effect of providing primary care patients with free and convenient access to a set of essential medicines. Half of the participants will receive free and convenient access to these essential medicines, while the other half will have usual access to medicines.

DETAILED DESCRIPTION:
Medication adherence is one important determinant of health outcomes. Approximately one half of treatments for chronic disease are not taken as directed. Cost is one of several important causes of poor adherence and it is particularly important for vulnerable people.

The size of many formularies makes it difficult for clinicians to know the safest and most effective medications to prescribe. This may partially explain poor medication selection. Short lists of essential medications have improved the the quality of prescribing.

ELIGIBILITY:
Inclusion Criteria:

* Cost related medicine non-adherence during last 12 months

Exclusion Criteria:

* Family member living at same address of patient who is already enrolled in this trial
* Patient joined practice during last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 784 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Appropriate medicine adherence | During entire study period (24 months)
  The percentage of patients taking medicines that are both (1) appropriate based on explicit criteria and (2) taken as prescribed or adhered to for 80 % of doses

SECONDARY OUTCOMES:
Percentage (%) of prescriptions that are appropriate. | During entire study period (24 months)
Percentage (%) of prescriptions that are adhered to. | During entire study period (24 months)
Hemoglobin A1c levels in patients with diabetes (adjusted for baseline) | Assessed between months 21 and 24 inclusive
Blood pressure in hypertensive patients (adjusted for baseline) | Assessed between months 21 and 24 inclusive
LDL cholesterol levels in patients taking a statin (adjusted for baseline | Assessed between months 21 and 24 inclusive
Healthcare costs including medication costs | During entire study period (24 months)

OTHER OUTCOMES:
Count of healthcare encounters | During entire study period (24 months)
  Includes ambulatory visits, emergency department visits, hospital admission, investigations and other healthcare utilization.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Municipality of Assiginack Family Health Team, Assiginack, Ontario
  - Huron Shores Family Health Team, Blind River, Ontario
  - St Michael's Hospital Academic Family Health Team, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available at the time of study completion.

REFERENCES:
- [Derived] Persaud N, Bedard M, Boozary A, Glazier RH, Gomes T, Hwang SW, Juni P, Law MR, Mamdani M, Manns B, Martin D, Morgan SG, Oh P, Pinto AD, Shah BR, Sullivan F, Umali N, Thorpe KE, Tu K, Wu F, Laupacis A; CLEAN Meds study team. Effect of Free Medicine Distribution on Health Care Costs in Canada Over 3 Years: A Secondary Analysis of the CLEAN Meds Randomized Clinical Trial. JAMA Health Forum. 2023 May 5;4(5):e231127. doi: 10.1001/jamahealthforum.2023.1127. PMID 37234014
- [Derived] Hess M, Wang R, Workentin A, Woods H, Persaud N. Effect of free medicine distribution on ability to make ends meet: post hoc quantitative subgroup analysis and qualitative thematic analysis. BMJ Open. 2022 Dec 22;12(12):e061726. doi: 10.1136/bmjopen-2022-061726. PMID 36549740
- [Derived] Persaud N, Bedard M, Boozary A, Glazier RH, Gomes T, Hwang SW, Juni P, Law MR, Mamdani M, Manns B, Martin D, Morgan SG, Oh P, Pinto AD, Shah BR, Sullivan F, Umali N, Thorpe KE, Tu K, Laupacis A; Carefully seLected and Easily Accessible at No Charge Medications (CLEAN Meds) study team. Adherence at 2 years with distribution of essential medicines at no charge: The CLEAN Meds randomized clinical trial. PLoS Med. 2021 May 21;18(5):e1003590. doi: 10.1371/journal.pmed.1003590. eCollection 2021 May. PMID 34019540
- [Derived] Charles O, Woods H, Ally M, Manns B, Shah BR, Wang R, Persaud N. Effect of free distribution of medicines on the process of care for adult patients with type 1 and type 2 diabetes and hypertension: post hoc analysis of randomised controlled trial findings. BMJ Open. 2021 Mar 15;11(3):e042046. doi: 10.1136/bmjopen-2020-042046. PMID 33722866
- [Derived] Yaphe H, Adekoya I, Steiner L, Maraj D, O'Campo P, Persaud N. Exploring the experiences of people in Ontario, Canada who have trouble affording medicines: a qualitative concept mapping study. BMJ Open. 2019 Dec 29;9(12):e033933. doi: 10.1136/bmjopen-2019-033933. PMID 31888944
- [Derived] Persaud N, Bedard M, Boozary AS, Glazier RH, Gomes T, Hwang SW, Juni P, Law MR, Mamdani MM, Manns BJ, Martin D, Morgan SG, Oh PI, Pinto AD, Shah BR, Sullivan F, Umali N, Thorpe KE, Tu K, Laupacis A; Carefully Selected and Easily Accessible at No Charge Medicines (CLEAN Meds) Study Team. Effect on Treatment Adherence of Distributing Essential Medicines at No Charge: The CLEAN Meds Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):27-34. doi: 10.1001/jamainternmed.2019.4472. PMID 31589276
- [Derived] Persaud N, Lee T, Ahmad H, Li W, Taglione MS, Rajakulasingam Y, Umali N, Boozary A, Glazier RH, Gomes T, Hwang SW, Juni P, Law M, Mamdani MM, Manns B, Martin D, Morgan S, Oh P, Pinto AD, Shah BR, Sullivan FM, Thorpe KE, Tu K, Laupacis A. Protocol for a randomised controlled trial evaluating the effects of providing essential medicines at no charge: the Carefully seLected and Easily Accessible at No Charge Medicines (CLEAN Meds) trial. BMJ Open. 2017 Jun 12;7(5):e015686. doi: 10.1136/bmjopen-2016-015686. PMID 28611089